CLINICAL TRIAL: NCT02687126
Title: Ultrasound Guided Technique for Internal Jugular Central Venous Catheterization in Pediatric Cardiac Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Gangalal National Heart Centre (Other)
Responsible Party: Principal Investigator, Santosh Sharma Parajuli, Doctor, Shahid Gangalal National Heart Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SGNHC
Record Dates: First submitted 2016-01-15; First posted 2016-02-22 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Accidental Puncture of Artery During Catheter Insertion
MeSH Terms: interventions — Catheterization, Central Venous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pediatric Cardiac Surgical Patients (Other): Central Venous Catheterization
  Interventions: Device: Central Venous Catheterization

INTERVENTIONS:
Device: Central Venous Catheterization — Ultrasound guided internal jugular venous catheterization

SUMMARY:
The purpose of the study is to evaluate the success rate using ultrasound as guidance during central venous cannulation in pediatric cardiac surgical patients.

DETAILED DESCRIPTION:
Central venous access may be essential in pediatric patients for fluid and a blood product administration, medication, parenteral nutrition, renal replacement therapy and hemodynamic monitoring. Obtaining central venous access in pediatric patients can be challenging, failure rates in pediatric patients range from 5% to 19% with reported complication rates from 2.5% to 22%. The landmark technique has been standard approach for many years. In comparison with landmark method, in pediatric patients, the use of ultrasound is associated with an increased success rate decreased operative time, reduced number of cannulation attempts , and a decreased number of carotid artery punctures. This study is designed to evaluate the success rate, complications, time taken for successful cannulation and their correlation with cross sectional area of the vein.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring central venous catheterization for elective cardiac surgery.
2. Age below 15 years.

Exclusion Criteria:

1. Patient's guardian's refusal
2. Bleeding disorders
3. Clotting abnormalities (platelets count < 75,000/cumm, INR > 2)
4. Local site of infection
5. Underlying pneumothorax, pleural effusion or preoperative insertion of chest tube

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santosh S Parajuli, MD, Principal Investigator — Shahid Gangalal National Heart Centre
Locations (1):
- Shahid Gangalal NationalHeart Centre, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Froehlich CD, Rigby MR, Rosenberg ES, Li R, Roerig PL, Easley KA, Stockwell JA. Ultrasound-guided central venous catheter placement decreases complications and decreases placement attempts compared with the landmark technique in patients in a pediatric intensive care unit. Crit Care Med. 2009 Mar;37(3):1090-6. doi: 10.1097/CCM.0b013e31819b570e. PMID 19237922
- [Result] Wigmore TJ, Smythe JF, Hacking MB, Raobaikady R, MacCallum NS. Effect of the implementation of NICE guidelines for ultrasound guidance on the complication rates associated with central venous catheter placement in patients presenting for routine surgery in a tertiary referral centre. Br J Anaesth. 2007 Nov;99(5):662-5. doi: 10.1093/bja/aem262. Epub 2007 Sep 14. PMID 17872936

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound Guided Central Venous Catheterization: Six month study of ultrasound guided internal jugular venous catheterization in pediatric cardiac surgical patients
Period: Data Collection
Arm/Group | Ultrasound Guided Central Venous Catheterization
Started | 106
Completed | 106
Not Completed | 0
Period: Data Analysis
Arm/Group | Ultrasound Guided Central Venous Catheterization
Started | 106
Completed | 106
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Demographic Variables: gender, age, weight, height, cross sectional area, body surface area
Arm/Group | Demographic Variables
Number analyzed (Participants) | 106
Age, Continuous [Median (Full Range); unit: Months] | 60 [1.5 to 180]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 41
Height [Median (Full Range); unit: Centimeters] | 102 [51 to 163]
Weight [Median (Full Range); unit: Kilograms] | 15 [3 to 54]
Body surface area [Median (Full Range); unit: Square of meter] — Body surface area was calculated using Mosteller's formula
  Square of meter | 0.655 [0.22 to 1.52]
Cross sectional area of the Internal Jugular Vein [Median (Full Range); unit: Square of centimeter] | 0.775 [0.12 to 2.01]

OUTCOME MEASURES:

1. Primary Outcome: Number of Attempts for Successful Central Venous Cannulation
Description: An attempt will be considered when complete withdrawal of the puncturing needle out of skin surface will occur
Time Frame: up to 24 hours after intervention
Measure: Mean (Standard Deviation); unit: Attempts
Groups:
- Number of Attempts: An attempt is considered unsuccessful if complete withdrawal of the puncture needle out of skin occurs
Arm/Group | Number of Attempts
Number analyzed (Participants) | 106
Attempts | 1.29 (0.59)

2. Secondary Outcome: Time to Successful Cannulation
Description: Time from skin prick to blood aspiration via the catheter immediately following the guide-wire removal
Time Frame: up to 1 hour after intervention
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Time to Successful Cannulation: Time taken in seconds from skin prick to aspiration of blood from catheter
Arm/Group | Time to Successful Cannulation
Number analyzed (Participants) | 106
Seconds | 134.06 (81.59)

3. Secondary Outcome: Number of Patients With Complications
Description: Arterial puncture, Hemothorax, Pneumothorax, Local site hematoma
Time Frame: up to 24 hours after intervention
Measure: Count of Participants; unit: Participants
Groups:
- Number of Complications: Complications were defined as arterial puncture, hemothorax, pneumothorax and local site hematoma
Arm/Group | Number of Complications
Number analyzed (Participants) | 106
Participants | 11

4. Other Pre Specified Outcome: Cross Sectional Area of Internal Jugular Vein
Description: Correlation of cross sectional area of internal jugular vein with number of attempts, time taken for successful cannulation and complication rate
Time Frame: up to 1 hour before intervention
Measure: Number; unit: Pearson's correlation Coefficient
Groups:
- Correlation: Correlation of cross sectional area of internal jugular vein with number of attempts, time taken for successful cannulation and complication rate
Arm/Group | Correlation
Number analyzed (Participants) | 106
Pearson's correlation Coefficient
  Number of attempts | -0.192
  Time for successful cannulation | -0.35
  Overall complications | 0.095

ADVERSE EVENTS:
Arm/Group | Number of Complications
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 11/106
Other Adverse Events (participants affected / at risk) | 11/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Complications (N=106)
Arterial puncture (Blood and lymphatic system disorders) | 11 (11)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Complications (N=106)
Local site hematoma (Skin and subcutaneous tissue disorders) | 11 (11)

LIMITATIONS AND CAVEATS:
Disease conditions of the patients may affect the size of the internal jugular vein. We did not evaluate the outcome variables in different disease conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes